CLINICAL TRIAL: NCT05573243
Title: Long-term Clinical Evaluation of Composite Restoration Using Two-steps Universal Adhesive in Non-carious Cervical Lesion: a Randomized Clinical Trial
Brief Title: Clinical Evaluation of Composite Restorations Using Two-steps Universal Adhesive in Non-carious Cervical Lesion (NCCL)
Acronym: NCCL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pipop Saikaew, Asst. Prof. Pipop Saikaew, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/DT086
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Non-carious Cervical Lesion
Keywords: clinical trial; universal adhesive; etch-and-rinse; selective enamel etching; self-etch

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Etch-and-rinse (Experimental): G2 Bond Universal bonded to NCCL using etch-and-rinse technique
  Interventions: Other: bonding strategies
- Selective enamel etching (Experimental): G2 Bond Universal bonded to NCCL using selective enamel etching technique
  Interventions: Other: bonding strategies
- self-etch (Experimental): G2 Bond Universal bonded to NCCL using self-etch technique
  Interventions: Other: bonding strategies

INTERVENTIONS:
Other: bonding strategies — The universal adhesive can be bonded using 3 different bonding strategies. Therefore, three bonding strategies will be assigned for 3 arms: etch-and-rinse, selective enamel etching, self-etch

SUMMARY:
The goal of this clinical study is to compare the clinical performance of a new 2-steps universal adhesive in patients with non-carious cervical lesions. The main question it aims to answer is: Is there any difference in clinical performance of a new 2-steps universal adhesives bonded with different etching strategies.

Participants will have restorations using a new 2-steps universal adhesives in different etching strategies.

* etch-and-rinse
* selective enamel etching
* self-etch

ELIGIBILITY:
Inclusion Criteria:

* Available for follow-up visits
* Have at least 28 teeth/ 20 teeth under occlusion
* Have at least 3 non-carious cervical lesions without peri-apical lesion. The lesion is not nearly exposed pulp and no history of previous restoration.

Exclusion Criteria:

* Rampant / uncontrolled caries
* Advanced untreated periodontal disease
* >2 cigarette packs/day
* Systemic or local disorders that could not undergo dental procedures
* Xerostomia
* Severe bruxism, clenching, TMD
* Pregnancy at the time of screening
* Known history of sensitivity to resin or related materials
* Fixed orthodontic appliance or planning to have orthodontic treatment within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity (modified USPHS) | 3 years
  tooth sensitivity to hot/cold water, tactile
retention (modified USPHS) | 3 years
  retention rate of the restoration that retain in the mouth after treatment
secondary caries (modified USPHS) | 3 years
  caries recurrent rate after restoration

SECONDARY OUTCOMES:
marginal adaptation (modified USPHS) | 3 years
  the quality of the restoration margin

CONTACTS AND LOCATIONS:
Overall Officials: Pipop Saikaew, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Dentistry, Manidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Paris Matos T, Perdigao J, de Paula E, Coppla F, Hass V, Scheffer RF, Reis A, Loguercio AD. Five-year clinical evaluation of a universal adhesive: A randomized double-blind trial. Dent Mater. 2020 Nov;36(11):1474-1485. doi: 10.1016/j.dental.2020.08.007. Epub 2020 Sep 12. PMID 32933775